CLINICAL TRIAL: NCT03225313
Title: Ultra Sound Guided Rectus Sheath Block or Field Block for Midline Hernia Repair: A Comparative Study
Brief Title: Comparison Between Ultra Sound Guided Rectus Sheath Block and Field Block for Midline Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Mohamed Hussein, Lecturer of Anesthesia and Surgical intensive care, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 722014
Record Dates: First submitted 2017-06-10; First posted 2017-07-21 (Actual); Results first posted 2019-07-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Ultrasound Guided Rectus Sheath Block; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Placebo Comparator): normal saline will be injected in the rectus sheath
  Interventions: Drug: Normal Saline Flush, 0.9% Injectable Solution_#5
- Rectus block group (Active Comparator): bupivicaine will be injected in the rectus sheath
  Interventions: Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#4
- Field block group (Experimental): bupivicaine will be injected locally in a circular fashion surrounding the site of the hernia
  Interventions: Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#4

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#4 — ultra sound guided injection into the rectus sheath
  Arms: Rectus block group
Drug: Normal Saline Flush, 0.9% Injectable Solution_#5 — injected into rectus sheath using ultrasound & locally surrounding the hernia
  Arms: control group
Drug: Bupivacaine Hydrochloride 0.5% Injection Solution_#4 — locally surrounding the hernia
  Arms: Field block group

SUMMARY:
Randomized double blinded controlled clinical trial will be done with a total number of 75 patients will be divided into 3 groups. To compare between Ultra-sound guided rectus sheath block VS Field block infiltration in providing a good analgesia for patients undergoing midline hernia repair to detect which one is superior.

DETAILED DESCRIPTION:
75 patients undergoing midline hernia repair under general anesthesia will be recruited and will be randomly allocated using closed envelope technique as follows: Control group, Local infilteration (Field block infilteration) group, Ultra sound Guided Rectus sheath block group.

General anesthesia will be standardized for all patients with :

2 µg kg-1 fentanyl and 2 mg kg-1 propofol. Neuromuscular blockade will be achieved with 0.5 mg kg-1 atracurium followed by tracheal intubation.

Muscle relaxation will be maintained by 0.1mg / kg / 30 minute of Atracrurium. Anesthesia will be maintained by sevoflurane. Mechanical ventilation will be adjusted with fresh gas flow oxygen in air 30-50% at a rate of 1 L min-1to maintain end-tidal carbon dioxide of 35-40 mm Hg and Spo2 greater than 94%.

BIS values will be maintained between 40 and 60. All surgical procedures will be done in the range between 10 am and 1 pm and by the same surgical team.

1. Control group : will receive field block using 0.3 ml/kg of normal saline at site of the hernia plus ultra- sound guided rectus sheath injection using 0.3 ml / kg of normal saline.
2. Field block group: will receive 0.3 ml / kg of 0.5% bupivicaine subcutaneously surrounding the site of the hernia following the induction of anesthesia and ultra-sound guided rectus sheath block with 0.3 ml / kg of normal saline.
3. Ultrasound guided rectus sheath block : Under sterile conditions a 21/22 G , 50- 100 milli meter length echogenic needle guided by the ultrasound into rectus sheath at the level of the umbilicus , using an - in plane technique. After -ve aspiration 0.3 ml/ kg of 0.5 % bupivicaine will be deposited on each side and the spread of local anesthesia will be observed by ultrasound plus 0.3 ml/kg of normal saline subcutaneously at the site of the hernia.

All solutions used will be prepared by a colleague who will not participate into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Elective midline hernia repair surgery.
2. Age: adult patients between 18 - 60 years old.
3. Gender: Both male and female.
4. ASA Class: I & II.

Exclusion Criteria:

1. Refusal of patient.
2. Pregnancy and lactation.
3. Fever or sepsis.
4. Patients ASA III or IV.
5. Addicts and drug abusers.
6. Patients taking corticosteroids or any cardio - active drugs.
7. Local infection at site of the injection.
8. Allergy to any of the study medications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: mohammed ma hussein, lecturer, Principal Investigator — Theodor Bilharz Research Institute
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ASA I & II patients. 25 patient in each group.
Pre-assignment Details: Prospective randomized double blinded controlled clinical trial was done with a total number of 75 patients divided into 3 groups .
Groups:
- Control Group: normal saline will be injected in the rectus sheath
  Normal saline: injected into rectus sheath & locally
- Ultra- Sound Rectus Sheath Block Group: bupivicaine will be injected in the rectus sheath
  Bupivacaine Hydrochloride: ultra sound guided injection into the rectus sheath
- Local Infilteration Group: bupivicaine will be injected locally
  Bupivacaine Hydrochloride: injected locally
Period: Overall Study
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Started | 25 (25 Patients) | 25 (25 Patients) | 25 (25 Patients)
Completed | 25 (25 Patients) | 25 (25 Patients) | 25 (25 Patients)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: count of participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 25 | 75
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.80 (9.941) | 42.20 (10.464) | 44.08 (8.544) | 43.76 (9.606)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 19 | 58
  Male | 3 | 8 | 6 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Egypt | 25 | 25 | 25 | 75
Body Weight in Kilograms [Mean (Standard Deviation); unit: Kilogram] | 82.7 (13.9) | 83.7 (11.8) | 82 (10.6) | 82.87 (12.115)

OUTCOME MEASURES:

1. Primary Outcome: Immediate Postoperative Pain
Description: Evaluation of the intensity of postoperative pain using Visual Analogue Scale (VAS) for pain: 0- 10 Scale; 0 the lowest pain score, 10 the highest pain scale.
  0 score: Better pain control achieved. 10 score: Worst pain control achieved. 3 score: Controllable pain control achieved.
Time Frame: evaluation of postoperative pain in patients immediately after the procedure.
Population: Evaluation of the intensity of postoperative pain using Visual Analogue Scale (VAS) for pain: 0- 10 Scale; 0 the lowest pain score, 10 the highest pain scale.
  0 score: Better pain control achieved. 10 score: Worst pain control achieved. 3 score: Controllable pain control achieved.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 7.36 (2.691) | 1.04 (1.837) | 6.56 (3.029)

2. Primary Outcome: Postoperative Pain at 2 Hours After Procedure.
Description: as for outcome 1
Time Frame: evaluation of postoperative pain in patients at 2 hours after procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 6.04 (1.645) | 1.20 (1.826) | 5.12 (1.833)

3. Primary Outcome: Postoperative Pain at 6 Hours After Procedure.
Description: as for outcome 1
Time Frame: Evaluation of postoperative pain in patients at 6 hours after procedure.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
score on a scale | 5.28 (2.011) | 2.64 (1.497) | 5.16 (2.304)

4. Secondary Outcome: Change in the Level of Serum Cortisol.
Description: Measurement of serum cortisol level (nmol/ liter) using the ELISA technique after 1 hour of the start of the surgery.
Time Frame: Measurement of serum cortisol level (nmol/ liter) using the ELISA technique after 1 hour of the start of the surgery.
Population: Measurement of serum cortisol level (nmol/ liter) using the ELISA technique after 1 hour of the start of the surgery.
Measure: Mean (Standard Deviation); unit: nmol/ liter
Groups:
- Rectus Block Group: bupivicaine will be injected in the rectus sheath
  Bupivacaine Hydrochloride: ultra sound guided injection into the rectus sheath
- Local Group: bupivicaine will be injected locally
  Bupivacaine Hydrochloride: injected locally
Arm/Group | Control Group | Rectus Block Group | Local Group
Number analyzed (Participants) | 25 | 25 | 25
nmol/ liter | 307.84 (220.569) | 214.00 (148.198) | 286.92 (225.404)

5. Secondary Outcome: Measurement of Serum Adrenaline Levels (ng/ml) Using ELISA Technique.
Description: Measurement of serum adrenaline levels (ng/ml) 1 hour after the start of the surgery using ELISA technique.
Time Frame: 1 hour after the start of the surgery using ELISA technique.
Population: Measurement of serum adrenaline levels (ng/ml) 1 hour after the start of the surgery using ELISA technique.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
ng/ml | 2.508 (1.2530) | 2.556 (1.4030) | 2.704 (1.1264)

6. Secondary Outcome: Measurement of Serum Noradrenaline Levels (ng/ml) Using ELISA Technique.
Description: Measurement of serum noradrenaline levels (ng/ml) 1 hour after the start of the surgery using ELISA technique.
Time Frame: 1 hour after the start of the surgery
Population: Measurement of serum noradrenaline levels (ng/ml) 1 hour after the start of the surgery using ELISA technique.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
ng/ml | 12.088 (4.6656) | 17.380 (9.0959) | 15.920 (7.3389)

7. Secondary Outcome: Measurement of Serum Cortisol Level (Nmol/ Liter) Using ELISA Technique.
Description: Measurement of serum cortisol level (nmol/ liter) using ELISA technique 30 minutes before the start of the surgery
Time Frame: 30 minutes before the start of the surgery
Population: Measurement of serum cortisol level (nmol/ liter) using ELISA technique 30 minutes before the start of the surgery
Measure: Mean (Standard Deviation); unit: nmol/ liter
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
nmol/ liter | 159.02 (119.455) | 327.05 (215.569) | 170.52 (91.421)

8. Secondary Outcome: Measurement of Serum Adrenaline Level (ng/ml) Using ELISA Technique.
Description: Measurement of serum adrenaline level (ng/ml) using ELISA technique 30 minutes before the start of the surgery.
Time Frame: 30 minutes before the start of the surgery
Population: Measurement of serum adrenaline level (ng/ml) using ELISA technique 30 minutes before the start of the surgery.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
ng/ml | 1.42 (0.774) | 3.96 (2.262) | 2.00 (1.416)

9. Secondary Outcome: Measurement of Serum Noradrenaline Levels (ng/ml) Using ELISA Technique.
Description: Measurement of serum noradrenaline levels (ng/ml) using ELISA technique 30 minutes before the start of the surgery.
Time Frame: 30 minutes before the start of the surgery.
Population: Measurement of serum noradreline levels (ng/ml) using ELISA technique 30 minutes before the start of the surgery.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
Number analyzed (Participants) | 25 | 25 | 25
ng/ml | 9.960 (4.2880) | 20.880 (10.5235) | 12.932 (6.4223)

ADVERSE EVENTS:
Time Frame: 24 hours after giving the local anaesthesia
Description: Cardiac arrhythmia.
Arm/Group | Control Group | Ultra- Sound Rectus Sheath Block Group | Local Infilteration Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT03225313/Prot_SAP_000.pdf